CLINICAL TRIAL: NCT00561054
Title: Open-Label, Uncontrolled, Multicenter, Phase II Study Evaluating the Efficacy and Safety of Cetuximab in Combination With Cisplatin & Gemcitabine as First-Line Therapy in Patients With Advanced Non Small Cell Lung Cancer
Brief Title: Efficacy and Safety of Cetuximab in Combination With Cisplatin Gemcitabine as First-Line Therapy in Advanced NSCLC
Acronym: Coimbra
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Portugues de Estudo do Cancro do Pulmao (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-000537-35
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Coimbra; NSCLC; CETUXIMAB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): CISPLATIN gENCITABINE cETUXIMAB
  Interventions: Drug: CETUXIMAB

INTERVENTIONS:
Drug: CETUXIMAB — 400 mg/m2 starting dose, 250 mg/m2 weekly dose

SUMMARY:
Lung cancer is the leading cause of cancer deaths worldwide. It is estimated that, in 2004, 173,700 new cases of lung cancer will be diagnosed in the United States alone and 164,440 deaths due to this disease will occur(13) . NSCLC accounts for approximately 80% of all lung cancers. Among NSCLC cases approximately 30% present with locally advanced and 40% with metastatic disease (14,15) . In metastatic disease, chemotherapy is the treatment of choice, but benefits obtained in survival have been modest. Five-year survival is less than 15%, probably due to diagnosis at late stages. Surgical results in earlier stages are poor compared to other tumor types (about 40% of recurrence in stages I-II). Results of chemotherapy in advanced stages are also poor (one-year survival of 40%) (15,17). It is commonly accepted that the standard treatment for advanced disease (stage IV and IIIb with malignant pleural effusion) consists of platinum-based chemotherapy(15,16) . However, there are many open questions in the management of these patients, such as the role of 3-drugs combinations, non-platinum-based therapies, and new biologic therapeutics' approaches. Currently, in the treatment of advanced NSCLC response rates of about 20%-30% and median survival times of 6 to 11 months have been achieved (16, 17, 18, 19, 20, 21, 22,). Several combinations of drugs are used and show similar efficacy. Cisplatin plus vinorelbine or Cisplatin plus Gemcitabine are among the most commonly used regimens in the first-line therapy of NSCLC.

DETAILED DESCRIPTION:
Criteria for inclusion Signed written informed consent Male or female ≥18 years of age Cito-histological diagnosis of NSCLC, stage IV Performance Status = 0 or 1 Measurable disease on CT scan - RECIST criteria White blood count ≥ 3 x 109/L, Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL Bilirubin level either normal or ≤1.5 x ULN ASAT and ALAT ≤ 2.5 x ULN (or 5 x ULN in case of liver metastases) Alkaline phosphatase ≤ 2,5 x ULN or ≤ 5 x ULN in case of bone metastases Creatinine clearance ≥ 50 ml/min Negative pregnancy test within one week before treatment start, if applicable Life expectancy of ≥ 3 months Availability of tumor sample (or able and willing to provide tumor sample) for EGFR assessment Effective contraception for both male and female patients if the risk of conception exists Criteria for exclusion Documented or symptomatic brain metastases Previous chemotherapy for NSCLC including adjuvant chemotherapy Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol Any investigational agent(s) within 4 weeks prior to entry Major surgery within 4 weeks prior to study entry Prior chest irradiation within 12 weeks prior to study entry (palliative radiation of bone lesions is allowed) Superior vena cava syndrome contra-indicating hydratation Previous exposure to EGF, monoclonal antibodies, signal transduction inhibitors or EGFR targeting therapy Myocardial infraction within 6 months prior to study entry, uncontrolled congestive heart failure; or any current grade 3 or 4 cardio-vascular disorder despite treatment Known allergic / hypersensitivity reaction to any of the components of study treatments Known drug abuse/ alcohol abuse Legal incapacity or limited legal capacity Symptomatic peripheral neuropathy (NCI-CTC) ≥ 2 and/or ototoxicity grade ≥ 2 , except if due to trauma or mechanical impairment due to tumor mass Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent Pregnancy or breastfeeding Any previous or concurrent malignancy other than nonmelanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for > 5 years will be allowed to enter the trial)

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female ≥18 years of age
* Cito-histological diagnosis of NSCLC, stage IV
* Performance Status = 0 or 1
* Measurable disease on CT scan - RECIST criteria
* White blood count ≥ 3 x 109/L, Neutrophils ≥ 1.5 x 109/L,
* platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL
* Bilirubin level either normal or ≤1.5 x ULN
* ASAT and ALAT ≤ 2.5 x ULN (or 5 x ULN in case of liver metastases)
* Alkaline phosphatase ≤ 2,5 x ULN or ≤ 5 x ULN in case of bone metastases
* Creatinine clearance ≥ 50 ml/min
* Negative pregnancy test within one week before treatment start, if applicable
* Life expectancy of ≥ 3 months
* Availability of tumor sample (or able and willing to provide tumor sample) for EGFR assessment
* Effective contraception for both male and female patients if the risk of conception exists

Exclusion Criteria:

* Documented or symptomatic brain metastases
* Previous chemotherapy for NSCLC including adjuvant chemotherapy
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to entry
* Major surgery within 4 weeks prior to study entry
* Prior chest irradiation within 12 weeks prior to study entry (palliative radiation of bone lesions is allowed)
* Superior vena cava syndrome contra-indicating hydratation
* Previous exposure to EGF, monoclonal antibodies, signal transduction inhibitors or EGFR targeting therapy
* Myocardial infraction within 6 months prior to study entry, uncontrolled congestive heart failure; or any current grade 3 or 4 cardio-vascular disorder despite treatment
* Known allergic / hypersensitivity reaction to any of the components of study treatments
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Symptomatic peripheral neuropathy (NCI-CTC) ≥ 2 and/or ototoxicity grade ≥ 2 , except if due to trauma or mechanical impairment due to tumor mass
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Pregnancy or breastfeeding
* Any previous or concurrent malignancy other than nonmelanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for > 5 years will be allowed to enter the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
oVERALL RESPONSE RATE | 30/11/2009

SECONDARY OUTCOMES:
tIME TO PROGRESSION oVERALL SORVIVAL SAFETY | 30/11/2009

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Barata, MD, Principal Investigator — Grupo Portugues de Estudo do Cancro do Pulmao
Locations (1):
- fERNANDO bARATA, Coimbra, Coimbra District, Portugal